CLINICAL TRIAL: NCT06348693
Title: Strategies for the Development of Multimodal Therapies in Tumors of the Central Nervous System: Identification of New Molecular and Metabolic Targets Implicated in Survival and Chemoresistance Involving Endothelial and Cancer Stem Cells
Brief Title: Development of Therapeutic Approaches Modulating Molecular Targets Implicated on Cancer Stem Cell-related Aggressiveness
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Other Study IDs: Gliotherapy
Record Dates: First submitted 2024-03-21; First posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-03

CONDITIONS: Glioblastoma; Glioma; Glioma Glioblastoma Multiforme
Keywords: cancer stem cells; tumor endothelial cells; sphingolipids; sphingosine-1-phosphate; platelets; biomarkers
MeSH Terms: conditions — Glioblastoma; Glioma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — cells from tumor biospsies and blood circulation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Glioma: Patients affected by brain tumors undergoing surgical resection; hypomethylation or hypermethylation of MGMT assessed post-surgery for patients affected by GBM; adult patients (≥18 years), both sexes; Patients undergoing Stupp protocol including patients aged > 70 years performing the hypofractionated protocol and three weeks of chemotherapy; Karnofsky Performance Status (KPS)> 60 assessed post-surgery; freely given written informed consent prior to any activity related to the study.
  Interventions: Other: cell isolation from tumor biopsies and biomarker investigation

INTERVENTIONS:
Other: cell isolation from tumor biopsies and biomarker investigation — cellular and molecular analysis on cancer stem cells and endothelial cells from tumor biopsies and investigation of tissue and systemic biomarkers

SUMMARY:
Tumors of the central nervous system affect 21 people per 100,000 every year, a figure that refers to countries with advanced economies, with an increase in incidence over time. Experimental evidence suggests that cancer stem cells (CSCs) may play a key role in the malignancy of these tumors. In fact, due to the hypoxic tumor microenvironment, these cells are able to create compensatory pathways that confer stem-like, angiogenic and pro-tumoral functions. Furthermore, it has been demonstrated that brain tumor stem cells are radio- and chemo-resistant and therefore not treatable with the therapeutic protocols currently in use. To date, in fact, there are no definitive treatments for the eradication of brain tumors. In this scenario, sphingolips, a class of lipid deputized to several physiological functions, are also involved in tumor onset, progression, drug resistance, and aggressiveness. In hypoxic tumor microenvironment, CSCs present a modified rheostat in the metabolism of sphingolipid, in favor of Sphingosine-1-phosphate (S1P).

S1P is an intermediate of sphingolipid metabolism, formed from sphingosine through the action of sphingosine kinases (SK). Increasing evidence suggests that S1P acts as a tumor-promoting signal, predominantly in the extracellular environment, regulating important cellular properties correlated with tumor potential.

The project aims to identify new molecular and metabolic targets involved in the survival and chemo-resistance of tumor stem cells in relation to the tumor microenvironment.

DETAILED DESCRIPTION:
Tumors of the central nervous system affect 21 people per 100,000 every year, a figure that refers to countries with advanced economies, with an increase in incidence over time. Among tumors of the central nervous system, Glioblastoma (GBM) is the most frequent and aggressive malignant tumor with an average life expectancy of approximately 12 months and a survival of less than 5% in the following 5 years to the diagnosis. The growth and progression of GBM are dependent on a specialized subpopulation of tumor cells called "cancer stem cells" (CSCs). CSCs are chemo- and radio-resistant, are responsible for relapses and therefore should constitute an important target of therapeutic strategies, but the mechanisms underlying their biology are still poorly understood. Hypoxia, through the hypoxia-inducible factor (HIF) and sphingolipid pathway, plays a key role in the control of tumor growth and angiogenesis and represents, perhaps, the most effective adaptation mechanism of the tumor itself. Indeed, The hypoxic microenvironment of solid tumors gives them greater aggressiveness, an increase in the expression of proteins linked to angiogenesis, anaerobic energy metabolism and adaptation to oxidative stress which facilitates the onset and proliferation of CSCs.

This study supports the evidence that the hypoxic microenvironment regulates the state of CSCs, and therefore influencing the response to the current pharmacological treatments.

Although S1P can act as an intracellular second messenger, most of its effects are exerted as an extracellular mediator, through binding to specific G protein-coupled receptors, originally known as EDGs and now called S1P receptors (S1PRs). Our group has previously demonstrated that acquired modifications in the metabolism of sphingolipids, in particular in the regulation of S1P, are able to confer stem-like and chemo-resistance properties to CSCs in patients with GBM.

The project aims to identify new molecular and metabolic targets involved in the survival and chemo-resistance of tumor stem cells in relation to the tumor microenvironment.

Through the study of sphingolipid metabolism, new markers and inhibitors will be identified to be delivered to inhibit CSC proliferation and tumor progression.

With this approach the investigators will be able to evaluate how the tumor microenvironment and the molecular and metabolic characteristics of the tumor influence cellular communication and whether this process can be influenced by new pharmacological treatments. This study could highlight new pathways and tumor-specific alterations to stratify new therapeutic strategies and to identify new potential biomarkers in diagnosis and monitoring, thus improving the prognosis of patients suffering from brain tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with glioma diagnosed histologically confirmed (WHO) undergoing surgical resection;
* hypomethylation or hypermethylation of MGMT assessed post-surgery for patients affected by GBM;
* adult patients (≥18 years), both sexes;
* Patients undergoing Stupp protocol including patients aged > 70 years performing the hypofractionated protocol and three weeks of chemotherapy;
* Karnofsky Performance Status (KPS)> 60 assessed post-surgery;
* freely given written informed consent prior to any activity related to the study. erine

Exclusion Criteria:

* patients who do not sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Considering the high heterogeneity of gliomas in relation to age, sex, surgical radicality, WHO performance status, MGMT methylation, molecular and biochemical characteristics, to demonstrate a benefit of the treatments that will be administered to stem and endothelial cells it will be necessary to consider a high sample size to allow for adequate subgroup analysis and to generate reliable data. To this end, the investigators will begin the study by analyzing 400 subjects affected by glioma.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2017-04-19 (Actual); Primary Completion 2025-11-21 (Estimated); Study Completion 2025-11-21 (Estimated)

PRIMARY OUTCOMES:
Investigation of molecular and metabolic signature of cancer stem cells to assess specific markers related to gliomagenesis and cancerogenesis. | Through study completion, an average of 3 years
  Evaluation of prognostic and predictive role of molecular and metabolic markers of the tumor. Determination of gene and protein expression of a panel of markers related to stemness, angiogenesis/hypoxia, and sphingolipid signaling.

SECONDARY OUTCOMES:
Biomarker investigation | Through study completion, an average of 3 years
  Identification of new tissue and circulating biomarkers with predictive and prognostic significance
Cellular response to pharmacological treatments | Through study completion, an average of 3 years
  Investigation of cellular response following new treatments determined by molecular and metabolic specific signature; determination of a panel of markers differently expressed following pharmacological treatments; evaluation of the prognostic and predictive role of tumor marker expression

CONTACTS AND LOCATIONS:
Overall Officials: Marco Locatelli, MD, PhD, Study Director — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico; Giovanni Marfia, MD, PhD, Study Chair — Fondazione IRCCS Ca' Granda Osp. Maggiore Policlinico, Istituto di Medicina Aerospaziale di Milano-Aeronautica Militare; Stefania E Navone, PhD, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy

REFERENCES:
- [Background] Marfia G, Navone SE, Fanizzi C, Tabano S, Pesenti C, Abdel Hadi L, Franzini A, Caroli M, Miozzo M, Riboni L, Rampini P, Campanella R. Prognostic value of preoperative von Willebrand factor plasma levels in patients with Glioblastoma. Cancer Med. 2016 Aug;5(8):1783-90. doi: 10.1002/cam4.747. Epub 2016 May 28. PMID 27236861
- [Result] Navone SE, Guarnaccia L, Rizzaro MD, Begani L, Barilla E, Alotta G, Garzia E, Caroli M, Ampollini A, Violetti A, Gervasi N, Campanella R, Riboni L, Locatelli M, Marfia G. Role of Luteolin as Potential New Therapeutic Option for Patients with Glioblastoma through Regulation of Sphingolipid Rheostat. Int J Mol Sci. 2023 Dec 21;25(1):130. doi: 10.3390/ijms25010130. PMID 38203299
- [Result] Guarnaccia M, Guarnaccia L, La Cognata V, Navone SE, Campanella R, Ampollini A, Locatelli M, Miozzo M, Marfia G, Cavallaro S. A Targeted Next-Generation Sequencing Panel to Genotype Gliomas. Life (Basel). 2022 Jun 24;12(7):956. doi: 10.3390/life12070956. PMID 35888045
- [Result] Campanella R, Guarnaccia L, Caroli M, Zarino B, Carrabba G, La Verde N, Gaudino C, Rampini A, Luzzi S, Riboni L, Locatelli M, Navone SE, Marfia G. Personalized and translational approach for malignant brain tumors in the era of precision medicine: the strategic contribution of an experienced neurosurgery laboratory in a modern neurosurgery and neuro-oncology department. J Neurol Sci. 2020 Oct 15;417:117083. doi: 10.1016/j.jns.2020.117083. Epub 2020 Aug 6. PMID 32784071
- [Result] Riboni L, Abdel Hadi L, Navone SE, Guarnaccia L, Campanella R, Marfia G. Sphingosine-1-Phosphate in the Tumor Microenvironment: A Signaling Hub Regulating Cancer Hallmarks. Cells. 2020 Feb 1;9(2):337. doi: 10.3390/cells9020337. PMID 32024090
- [Result] Campanella R, Guarnaccia L, Cordiglieri C, Trombetta E, Caroli M, Carrabba G, La Verde N, Rampini P, Gaudino C, Costa A, Luzzi S, Mantovani G, Locatelli M, Riboni L, Navone SE, Marfia G. Tumor-Educated Platelets and Angiogenesis in Glioblastoma: Another Brick in the Wall for Novel Prognostic and Targetable Biomarkers, Changing the Vision from a Localized Tumor to a Systemic Pathology. Cells. 2020 Jan 25;9(2):294. doi: 10.3390/cells9020294. PMID 31991805
- [Result] Abdel Hadi L, Anelli V, Guarnaccia L, Navone S, Beretta M, Moccia F, Tringali C, Urechie V, Campanella R, Marfia G, Riboni L. A bidirectional crosstalk between glioblastoma and brain endothelial cells potentiates the angiogenic and proliferative signaling of sphingosine-1-phosphate in the glioblastoma microenvironment. Biochim Biophys Acta Mol Cell Biol Lipids. 2018 Oct;1863(10):1179-1192. doi: 10.1016/j.bbalip.2018.07.009. Epub 2018 Jul 26. PMID 30056170
- [Result] Marfia G, Campanella R, Navone SE, Di Vito C, Riccitelli E, Hadi LA, Bornati A, de Rezende G, Giussani P, Tringali C, Viani P, Rampini P, Alessandri G, Parati E, Riboni L. Autocrine/paracrine sphingosine-1-phosphate fuels proliferative and stemness qualities of glioblastoma stem cells. Glia. 2014 Dec;62(12):1968-81. doi: 10.1002/glia.22718. Epub 2014 Jul 5. PMID 25042636
- [Result] Navone SE, Marfia G, Invernici G, Cristini S, Nava S, Balbi S, Sangiorgi S, Ciusani E, Bosutti A, Alessandri G, Slevin M, Parati EA. Isolation and expansion of human and mouse brain microvascular endothelial cells. Nat Protoc. 2013 Sep;8(9):1680-93. doi: 10.1038/nprot.2013.107. Epub 2013 Aug 8. PMID 23928501
- See also: website Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico — https://www.policlinico.mi.it/reparti/40/neurochirurgia